CLINICAL TRIAL: NCT01424384
Title: Emotional Processing in Healthy Male Volunteers Treated With GSK424887. A Single Centre, Randomised, Double-blind, Placebo-controlled Parallel Group Study
Brief Title: Emotional Processing in Healthy Volunteers in the Presence of an Investigational Anxiolytic
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 105012
Record Dates: First submitted 2010-02-12; First posted 2011-08-29 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Depressive Disorder and Anxiety Disorders
Keywords: healthy volunteers; Anxiety Disorder; neuropsychological tests
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders | interventions — Citalopram; N-(1-(3-chloro-1-naphthalenyl)ethyl)-2-(4-(4-fluorophenyl)-1-methyl-4-piperidinyl)-N-methylacetamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Citalopram (Active Comparator): Marketed comparitor
  Interventions: Drug: Citalopram
- Investigational Medicinal Product (Experimental): GSK424887
  Interventions: Drug: GSK424887
- Placebo To Match Treatment (Placebo Comparator): Placebo control
  Interventions: Drug: Plactebo To Match

INTERVENTIONS:
Drug: Citalopram — Neurophysiological testing.
  Arms: Citalopram
Drug: GSK424887 — Neurophysiological testing
  Arms: Investigational Medicinal Product
Drug: Plactebo To Match — Neurophysiological testing
  Arms: Placebo To Match Treatment

SUMMARY:
This will be a phase I, single centre, randomised, double blind, double-dummy, placebo controlled, parallel group single-dose study in healthy volunteers. The purpose of this study is to assess the effect of a single-dose administration of GSK424887, a potent, selective competitive antagonist of the human Neurokinin 1 (NK1) receptor and a potent inhibitor of the human serotonin transporter (SERT), at the maximum dosage of 100 mg versus placebo and versus citalopram (20 mg) on emotional processing in healthy male volunteers. Pharmacokinetics and safety following oral administration of GSK424887 will be also evaluated. An Emotional Test Battery (ETB) previously used to characterise the effects of antidepressants on positive and negative emotion processing in Healthy Volunteers and patients will be used. We hypothesise that GSK424887 will modulate emotional information processing acutely. We anticipate that these effects may be manifest at sub-effective levels of NK1 and SERT receptor occupancy, thus providing pharmacodynamic evidence of the synergistic interaction of the two mechanisms in humans.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males with no neurological, or history of psychiatric illness
2. Aged between 18 and 45 years
3. Agree to use contraception
4. BMI range of 18 to 33 kg/m²
5. Fluent English speakers
6. Non smoker or light smoker

Exclusion Criteria:

1. Positive pre-study drug/alcohol screen or regular alcohol consumption
2. Positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
3. On prescription or non prescription drug
4. Exposure to more than four new chemical entities within 12 months prior to the first dosing day
5. Consumption of large amounts of caffeinated drinks
6. Significant hearing impairment
7. Previous experience of the emotional test battery experimental procedures

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2008-09-19 (Actual); Primary Completion 2009-04-30 (Actual); Study Completion 2009-04-30 (Actual)

PRIMARY OUTCOMES:
Multiple emotional and psychometric battery of tests | < 1 day
Adverse Events, laboratory values, vital signs, ECGs | < 1 day

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Harmer CJ, Dawson GR, Dourish CT, Favaron E, Parsons E, Fiore M, Zucchetto M, Bifone A, Poggesi I, Fernandes S, Alexander RC, Goodwin GM. Combined NK(1) antagonism and serotonin reuptake inhibition: effects on emotional processing in humans. J Psychopharmacol. 2013 May;27(5):435-43. doi: 10.1177/0269881112472558. Epub 2013 Feb 12. PMID 23407644
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 105012 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/105012?search=study&study_ids=105012#rs
- Available data/document: Study Protocol: 105012 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 105012 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 105012 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 105012 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 105012 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 105012 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 105012 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register